CLINICAL TRIAL: NCT01638598
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 1021958 in Healthy Chinese and Japanese Male Volunteers (Placebo-controlled, Randomised and Double-blind Within Dose Groups)
Brief Title: Single Rising Oral Doses of BI 1021958 in Healthy Chinese and Japanese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1310.3
Record Dates: First submitted 2012-07-02; First posted 2012-07-12 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — Drug Evaluation

ARMS (5):
- BI 1021958 dose group 1 (Experimental): subject to receive a tablet containing dose group 1 BI 1021958 single dose
  Interventions: Drug: Test drug; Drug: matching placebo
- BI 1021958 dose group 2 (Experimental): subject to receive a tablet containing dose group 2 BI 1021958 single dose
  Interventions: Drug: matching placebo; Drug: Test drug
- BI 1021958 dose group 3 (Experimental): subject to receive a tablet containing dose group 3 BI 1021958 single dose
  Interventions: Drug: Test drug; Drug: matching placebo
- BI 1021958 dose group 4 (Experimental): subject to receive a tablet containing dose group 4 BI 1021958 single dose
  Interventions: Drug: matching placebo; Drug: Test drug
- BI 1021958 dose group 5 (Experimental): subject to receive a tablet containing dose group 5 BI 1021958 single dose
  Interventions: Drug: Test drug; Drug: matching placebo

INTERVENTIONS:
Drug: matching placebo — matching placebo in each dose level
  Arms: BI 1021958 dose group 2
Drug: Test drug — BI 1021958
  Arms: BI 1021958 dose group 3
Drug: matching placebo — matching placebo in each dose level
  Arms: BI 1021958 dose group 4
Drug: Test drug — BI 1021958
  Arms: BI 1021958 dose group 2
Drug: Test drug — BI 1021958
  Arms: BI 1021958 dose group 5
Drug: Test drug — BI 1021958
  Arms: BI 1021958 dose group 1
Drug: Test drug — BI 1021958
  Arms: BI 1021958 dose group 4
Drug: matching placebo — matching placebo in each dose level
  Arms: BI 1021958 dose group 1
Drug: matching placebo — matching placebo in each dose level
  Arms: BI 1021958 dose group 3
Drug: matching placebo — matching placebo in each dose level
  Arms: BI 1021958 dose group 5

SUMMARY:
Safety,tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of BI 1021958 after single rising doses (SRD) in healthy Asian male volunteers

ELIGIBILITY:
Inclusion criteria:

1. Healthy males based upon a complete medical history, including a physical examination, vital signs (blood pressure, pulse rate), 12-lead ECG, and clinical laboratory tests
2. Chinese ethnicity, Japanese ethnicity according to the following criteria Japanese; born in Japan, be a current Japanese passport holder, have lived outside of Japan <5 years, and have parents and grandparents who were all born in Japan Chinese; ethnic Chinese, born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in China
3. Age within the range of 20 to 45 years
4. Body mass index within the range of 18.5 and 25 kg/m2
5. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion criteria:

1. Any finding of the medical examination (including Blood Pressure, Pulse Rate, ECG and Safety laboratory) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy/hypersensitivity to the study drug or its excipients)
9. Intake of drugs with a long half-life (more than 24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to administration
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval (based on the knowledge at the time of protocol preparation) within 10 days prior to administration
11. Participation in another trial with an investigational drug administration within 2 months prior to administration
12. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 30 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within 4 weeks prior to administration)
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of trial site
19. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval more than 450 ms), heart rate outside 45 to 90 bpm, or any other relevant ECG findings at screening
20. A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of long QT Syndrome)
21. Subjects considered unsuitable for inclusion by the investigator, e.g. because considered not able to understand and comply with study requirements, or have any condition which in the opinion of the investigator would not allow safe participation in the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The number (%) of subjects with related adverse events. | up to 17 days postdose

SECONDARY OUTCOMES:
AUC0-inf (area under the concentration-time curve of BI 1021958 in plasma over the time interval from 0 extrapolated to infinity) | up to day 4 postdose
AUC0-tz (area under the concentration-time curve of BI 1021958 in plasma over the time interval from 0 up to the last quantifiable data point) | up to day 4 postdose
AUC0-12 (area under the concentration-time curve of BI 1021958 in plasma over the time interval from the time point 0 until the time point 12 h) | up to day 4 postdose
Cmax (maximum measured concentration of BI 1021958 in plasma) | up to day 4 postdose
AUC0-24 (area under the concentration-time curve of BI 1021958 in plasma over the time interval from the time point 0 until the time point 24 h) | up to day 4 postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1310.3.8201 Boehringer Ingelheim Investigational Site, Seoul, South Korea